CLINICAL TRIAL: NCT06733610
Title: A Clinical Study Evaluating the Safety and Preliminary Efficacy of Universal Allogeneic CAR T-cell Therapy Targeting CD19 and BCMA in Patients with Autoimmune Hemolytic Anemia Have Failed ≥ 3 Lines of Therapy
Brief Title: CAR T-cell Therapy Targeting CD19 and BCMA in Patients with AIHA Who Have Failed ≥3 Lines of Therapy.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Xi'niao Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024096
Record Dates: First submitted 2024-12-06; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Hemolytic Anemia; CD19/BCMA CAR T-cells; Universal Allogeneic CAR T-cells
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UCAR T-cell group (Experimental): Universal allogeneic anti-CD19/BCMA CAR T-cells.
  Interventions: Biological: universal allogeneic anti-CD19/BCMA CAR T-cells

INTERVENTIONS:
Biological: universal allogeneic anti-CD19/BCMA CAR T-cells — A single injection of UCAR T-cells, referred to as universal allogeneic anti-CD19/BCMA CAR T-cells.

SUMMARY:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal allogeneic anti-CD19/BCMA CAR T-cells in AIHA who have failed ≥ 3 lines of therapy.

DETAILED DESCRIPTION:
This is an investigator-initiated trial to evaluate the safety and efficacy of universal allogeneic anti-CD19/BCMA CAR T-cells in autoimmune hemolytic anemia who have failed ≥ 3 lines of therapy.

Study intervention consists of a single infusion of universal allogeneic CAR T-cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

Interim analysis will be performed when participants finish the visit 12 weeks after CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Flow cytometry detected positive B cell CD19 or BCMA in the patient's peripheral blood.
* Patients diagnosed with AIHA, including warm antibody type, cold agglutinin disease, mixed type, and other types of AIHA, with diagnostic criteria referring to the "Chinese Adult Autoimmune Hemolytic Anemia Diagnosis and Treatment Guidelines (2023 Edition)"
* The definition of recurrent/refractory AIHA that has received at least 3 failed lines of treatment is symptomatic anemia (hemoglobin<100g/L) that persists after a routine treatment cycle of at least 6 months and is still ineffective or reappears after disease remission. The definition of conventional treatment: treatment with glucocorticoids and/or rituximab, as well as any 1-2 or more of the following immunomodulatory drugs: cyclophosphamide, azathioprine, mycophenolate mofetil, cyclosporine A, azathioprine, danazol, bendamustine, fludarabine, bortezomib, and biologics including daratumumab, BTK inhibitors, Syk inhibitors, and complement inhibitors.
* ECOG ≤ 2
* Functional requirements for major organs are as follows:

  1. . The bone marrow function needs to meet: a Neutrophil count ≥ 1.0 × 10 ^ 9/L; b. Platelets ≥ 30 × 10 ^ 9/L.
  2. Liver function: ALT ≤ 3 × UL; AST ≤ 3×ULN； Total bilirubin ≤ 2.0 × ULN (excluding Gilbert syndrome, total bilirubin ≤ 3.0 × ULN).
  3. Renal function: creatinine clearance rate (CrCl) ≥ 30 ml/min (Cockcroft/Gault formula, excluding acute CrCl decline caused by the disease itself).
* Female subjects of childbearing potential and male subjects with partners of childbearing potential must use medically approved contraception or abstinence during the study treatment period and for at least 6 months after the end of the study treatment; Female subjects of childbearing potential must have a negative Human chorionic gonadotropin (HCG) test within 7 days before study enrollment and not be lactating.
* Willing to participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Subjects with a history of severe drug allergies or allergic tendencies.
* Presence or suspicion of uncontrolled or treatment-required fungal, bacterial, viral, or other infections.
* Subjects with central nervous system diseases caused by autoimmune diseases or non-autoimmune diseases (including epilepsy, psychosis, organic brain syndrome, cerebral vascular accidents, encephalitis, central nervous system vasculitis).
* Subjects with insufficient cardiac function
* Subjects with congenital immunoglobulin deficiencies
* History of malignancy within five years
* Subjects with end-stage renal failure
* Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA >ULN; subjects positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA; individuals positive for human immunodeficiency virus (HIV) antibody; individuals positive for syphilis testing
* Subjects with psychiatric disorders and severe cognitive impairments
* Subjects who have used immunosuppressive agents or biologics with therapeutic effects on the disease within five half-life before enrollment
* Pregnant women or women planning to conceive
* Active infection, active rheumatic and immune disease, drug induced and diagnosed lymphoproliferative tumor associated secondary AIHA patients
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
The number and severity of dose-limiting toxicity (DLT) events | Within 28 Days After UCAR T-cell Infusion
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, and the ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells.
The total number, incidence, and severity of AEs | Up to 12 Months After UCAR T-cell Infusion
Clinical response of AIHA who have failed ≥ 3 lines of therapy | Up to 24 Weeks After UCAR T-cell Infusion
  Rates of CR, CRi, PR, ORR

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center and Red Blood Cell Disorders Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No